CLINICAL TRIAL: NCT05715762
Title: Determine the Effects of Prone Positioning and Nitric Oxide in Adult COVID-19 Patients With ARDS by Electrical Impedance Tomography
Brief Title: Determine the Effects of Prone Positioning and NO in COVID-19 ARDS by EIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: eit20221221
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Respiratory Distress Syndrome, Adult; COVID-19
Keywords: Respiratory Distress Syndrome; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Ventilation in supine position: Patients are ventilated in supine position.
- Ventilation in supine position and NO inhalation: Patients are ventilated in supine position with NO inhalation for 1 hour.
  Interventions: Drug: NO inhalation
- Ventilation in prone position for 1 hour: Patients are ventilated in prone position for 1 hour.
  Interventions: Behavioral: prone postion
- Ventilation in prone position for 2 hours plus NO inhalation for 1 hour: Patients are ventilated in prone position for 1 hour followed by ventilation in prone position with NO inhalation for 1 hour.
  Interventions: Behavioral: prone postion; Drug: NO inhalation
- Ventilation in prone position for 3 hours: Patients are ventilated in prone position for 1 hour followed by ventilation in prone position with NO inhalation for 1 hour. Then they are ventilated in prone position alone for 1 hour.
  Interventions: Behavioral: prone postion
- Ventilation in prone position for 16 hours: Patients are ventilated in prone position for 1 hour followed by ventilation in prone position with NO inhalation for 1 hour. Then they are ventilated in prone position alone for 14 hours.
  Interventions: Behavioral: prone postion
- Ventilation in re-supine position for 3 hours: Patients are ventilated in supine position for 3 hours followed by ventilation in prone position for 16 hours.

INTERVENTIONS:
Behavioral: prone postion — ventilation at prone positioning
  Other Names: PPV
  Groups: Ventilation in prone position for 1 hour; Ventilation in prone position for 16 hours; Ventilation in prone position for 2 hours plus NO inhalation for 1 hour; Ventilation in prone position for 3 hours
Drug: NO inhalation — NO inhalation at 20 ppm
  Groups: Ventilation in prone position for 2 hours plus NO inhalation for 1 hour; Ventilation in supine position and NO inhalation

SUMMARY:
We aims to investigate the effects of prone positioning and nitric oxide inhalation in adult patients who is diagnosed with COVID-19 associated acute respiratory distress syndrome by electrical impedance tomography.

DETAILED DESCRIPTION:
The investigators aim to investigate the effects of prone positioning and nitric oxide inhalation in adult patients who is diagnosed with COVID-19 associated acute respiratory distress syndrome by electrical impedance tomography (EIT).

The EIT assessment is performed in patients ventilated in supine position, supine position with NO inhalation for 1 hour, prone position for 1 hour, prone position for 2 hours with NO inhalation for 1 hour, prone position for 3 hours, prone position for 16 hours, re-supine position for 3 hours. Arterial blood gas (ABG) analysis results, ventilator parameters and hemodynamic parameters are also recorded at each time point.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who have COVID-19-associated acute respiratory distress syndrome

Exclusion Criteria:

* patients who refuse to participate in the study; unable to use EIT, such as open-chest surgery with chest tube placement; have contraindication for prone positioning, including pregnant, post-abdomen surgery within a week; hypercapnic respiratory failure.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients who have COVID-19-associated acute respiratory distress syndrome
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
oxygenation status | 1 day
  To evaluate the oxygenation parameters
regional distribution of pulmonary perfusion | 1 day
  To evaluate the effect of prone positon and NO inhalation on pulmonary blood flow distribution.
regional distribution of pulmonary ventilation | 1 day
  To evaluate the effect of prone positon and NO inhalation on pulmonary vetilation distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No